CLINICAL TRIAL: NCT02618226
Title: Diagnostic Accuracy of Optic Nerve Ultrasound for the Detection of Intracranial Hypertension and Prediction of Therapeutic Intensity Level and Mortality Following Severe Traumatic Brain Injury (ONUS-TBI): a Prospective Blinded Study
Brief Title: Optic Nerve Ultrasound in Severe Traumatic Injury
Acronym: ONUS-TBI
Status: Completed | Type: Observational
Sponsor: University of Michigan (Other)
Collaborators: All India Institute of Medical Sciences (Other); National Institutes of Health (NIH) (NIH); National Institute for Biomedical Imaging and Bioengineering (NIBIB) (NIH)
Responsible Party: Principal Investigator, Venkatakrishna Rajajee, Clinical Associate Professor, Neurosurgery and Neurology Medical Director, Neurointensive Care, University of Michigan
Other Study IDs: HUM00092614; IEC/NP-407/14.11.2014, RP (Other: All India Institute of Medical Sciences (AIIMS)); R03EB019352 (NIH)
Record Dates: First submitted 2015-11-19; First posted 2015-12-01 (Estimated); Last update posted 2021-01-05 (Actual); Status verified 2021-01

CONDITIONS: Traumatic Brain Injury; Intracranial Hypertension
Keywords: Traumatic Brain Injury; TBI; Optic nerve ultrasound; ONUS; Intracranial pressure; ICP; Intracranial hypertension
MeSH Terms: conditions — Brain Injuries, Traumatic; Intracranial Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Optic nerve ultrasound: Optic nerve sheath diameter (ONSD) measurement will be performed in subjects with concomitant measurement of Intracranial Pressure (ICP) from an invasive ICP monitor. The operator measuring ONSD will be blinded to concomitant ICP.
  Interventions: Device: Optic nerve ultrasound

INTERVENTIONS:
Device: Optic nerve ultrasound — Measurement of ONSD with concomitant invasive ICP measurement will be performed at enrollment and at least daily for a total of 7 days. Additional measurements of ONSD may be performed at any time following any decline in Glasgow Coma Scale (GCS) score by 2+ points during the 7 day period.

SUMMARY:
Prospective study of diagnostic accuracy of optic nerve sheath diameter measurement (index study) in traumatic brain injury with simultaneous invasive intracranial pressure monitoring as the reference standard.

DETAILED DESCRIPTION:
Background and Rationale:

Traumatic brain injury (TBI) is a public health problem of epidemic proportions both in the United States (US) and India. Trauma is estimated to be the leading cause of death in the age group 20-40 years in India and accounts for 2-3% loss of gross domestic product (GDP) every year. The incidence of TBI in India is among the highest in the world and is rapidly rising along with a rapid increase in automobile density. Compared to the United States, poor outcomes reported following TBI in India can be attributed to several factors including underdeveloped pre-hospital care, problems with transport to appropriate medical attention, limited availability of centers for trauma care, lack of appropriate training and expertise and lack of application of standards of TBI care widely accepted in the developed world. Over the last two decades the management of TBI in the US and Europe has centered on the guidelines developed by the Brain Trauma Foundation (BTF). Severe TBI, defined by a Glasgow Coma Scale <8, carries the worst prognosis, with a mortality of 30-40% in reports from India compared to 10-20% in the US. Monitoring of the Intracranial Pressure (ICP) is an integral part of the management of severe TBI, with the BTF recommending monitoring of ICP in appropriate candidates and maintenance of ICP at <20-25mmHg using a range of therapeutic options. The rationale for this recommendation lies in the fact that ICP>20mmHg is associated with clinical neurological decline and that Cerebral Perfusion Pressure [Mean Arterial Pressure (MAP) - ICP] <50mmHg is associated with worse neurological outcomes. Importantly, studies examining TBI have demonstrated an increase in 2-week mortality with non-use of ICP monitoring. Moreover adherence to guidelines on the management of ICP, including treatment of ICP>25mmHg, have been associated with a significant decline in mortality in New York state.

While widely accepted as the standard of care in the US, invasive ICP is not considered the standard of care in the developing world. Rather, clinical equipoise is considered to exist on the best way to measure ICP in these regions. A randomized controlled trial performed in Bolivia and Ecuador comparing an invasive ICP monitoring-based management protocol with a management protocol without invasive monitoring demonstrated no difference in neurological outcomes. While this trial may have been confounded by other, important differences between the interventions in both arms, it does illustrate the fact that invasive monitoring is not the current standard of care in the developing world. While the appropriate role and indications for invasive ICP monitoring in the developing world may be a matter of debate, the strong association between appropriate ICP management and mortality observed in other studies suggests that an urgent, unmet need exists for a low-cost, low-risk, non-invasive, point-of-care alternative to invasive monitoring for the detection of life-threatening increases in ICP following TBI. While the need for such a tool may be greatest in the developing world, where invasive monitoring is mostly unavailable, a validated non-invasive ICP monitor would also be of great value in the US, in potentially decreasing the risks of intracranial placement as well as the costs of invasive monitoring. While Optic Nerve Ultrasound (ONUS) is a promising noninvasive tool for the detection of life threatening intracranial hypertension, it is neither a continuous nor a quantitative measure of ICP and is unlikely to entirely replace invasive monitoring. The greatest potential value of a noninvasive diagnostic tool such as ONUS may be to function as a screening tool to permit early initiation of life-saving treatment measures and to decrease the burden of risk and expense associated with invasive monitoring. As a screening tool the sensitivity for the detection of intracranial hypertension will need to be high, while a moderate specificity may be acceptable, since a noninvasive measurement suggesting an increased likelihood of elevated ICP will likely lead to the placement of an invasive ICP monitor to follow the response to therapeutic intervention. Early identification of patients at risk of death from elevated ICP using noninvasive assessment tools may permit providers to both initiate treatment earlier and target limited resources toward these high-risk individuals.

Objective:

Aim 1: To determine the optimal optic nerve sheath diameter (ONSD) measurement for the detection of raised intracranial pressure (ICP) in Indian patients using Receiver Operating Characteristic (ROC) curves, with emphasis on a cut-off with high sensitivity and acceptable specificity, as appropriate for a screening tool.

Hypothesis- An ONSD threshold will be identified to maximize the true positive rate (>0.98) with acceptable specificity (>80%) for the detection of elevated ICP (>25mmHg).

Aim 2: To evaluate whether the optic nerve sheath diameter predicts Therapeutic Intensity Level, in-hospital mortality and discharge functional outcome following severe traumatic brain injury.

Hypothesis- The highest measured optic nerve sheath diameter within the first 48 hours in a patient with TBI will be associated with the Therapeutic Intensity Level, mortality during hospitalization and discharge functional outcome.

Study setting: The Jai Prakash Narayan Apex Trauma Center (JPNATC) at the All India Institute of Medical Sciences (AIIMS), New Delhi, is the apex referral center for TBI in New Delhi as well as from much of the rest of the country. It has 30 triage and 36 ICU beds, with 300-600 severe TBI admissions every year.

ELIGIBILITY:
Inclusion Criteria:

1. Adult (age>18 years) patients
2. Severe TBI (GCS<8)
3. First measurement feasible <48 hours from time of injury
4. Clinical decision has been made to place an invasive ICP monitor, based on the recommendations of the Brain Trauma Foundation.

I. GCS<8 and Abnormal CT brain OR II. GCS<8 and Normal CT brain PLUS any 2 of the following

1. Age>40
2. Systolic blood pressure<90
3. Unilateral or Bilateral Posturing

Exclusion Criteria:

1. Patient not expected to survive >48 hours from the time of enrollment
2. Known injury to the globe of the eye or the optic nerve
3. Therapeutic Intensity Level 3 or 4 attained before ONSD measurement can be performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe TBI in the neurotrauma ICU who meet inclusion/exclusion.
Sampling Method: Non-Probability Sample
Enrollment: 117 (Actual)
Dates: Start 2016-01; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Intracranial Pressure (ICP) >25mmHg | Days 1-7
  Accuracy of ONSD measurement (index test) compared to the reference standard- ICP>25mmHg on concomitant invasive monitoring

SECONDARY OUTCOMES:
Therapeutic Intensity Level (TIL) | Assessed at time of discharge from the neurotrauma intensive care unit- Average expected to be about 7 days
  Highest Therapeutic Intensity Level attained during the ICU admission
In-Hospital Mortality | At Discharge from inpatient admission- Average expected to be about 30 days
  All-cause mortality during the inpatient admission
Poor functional outcome at discharge- Glasgow Outcome Scale <4 | At Discharge from inpatient admission- Average expected to be about 30 days
  Moderate or low disability at the time of discharge

CONTACTS AND LOCATIONS:
Overall Officials: Venkatakrishna (Krishna) Rajajee, MD, Principal Investigator — University of Michigan
Locations (1):
- All India Institute of Medical Sciences (AIIMS), New Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Coronado VG, Xu L, Basavaraju SV, McGuire LC, Wald MM, Faul MD, Guzman BR, Hemphill JD; Centers for Disease Control and Prevention (CDC). Surveillance for traumatic brain injury-related deaths--United States, 1997-2007. MMWR Surveill Summ. 2011 May 6;60(5):1-32. PMID 21544045
- [Background] Langlois JA, Rutland-Brown W, Wald MM. The epidemiology and impact of traumatic brain injury: a brief overview. J Head Trauma Rehabil. 2006 Sep-Oct;21(5):375-8. doi: 10.1097/00001199-200609000-00001. PMID 16983222
- [Background] Gururaj G. Road traffic deaths, injuries and disabilities in India: current scenario. Natl Med J India. 2008 Jan-Feb;21(1):14-20. PMID 18472698
- [Background] Gururaj G. Epidemiology of traumatic brain injuries: Indian scenario. Neurol Res. 2002 Jan;24(1):24-8. doi: 10.1179/016164102101199503. PMID 11783750
- [Background] Brain Trauma Foundation; American Association of Neurological Surgeons; Congress of Neurological Surgeons; Joint Section on Neurotrauma and Critical Care, AANS/CNS; Bratton SL, Chestnut RM, Ghajar J, McConnell Hammond FF, Harris OA, Hartl R, Manley GT, Nemecek A, Newell DW, Rosenthal G, Schouten J, Shutter L, Timmons SD, Ullman JS, Videtta W, Wilberger JE, Wright DW. Guidelines for the management of severe traumatic brain injury. VI. Indications for intracranial pressure monitoring. J Neurotrauma. 2007;24 Suppl 1:S37-44. doi: 10.1089/neu.2007.9990. No abstract available. PMID 17511544
- [Background] Juul N, Morris GF, Marshall SB, Marshall LF. Intracranial hypertension and cerebral perfusion pressure: influence on neurological deterioration and outcome in severe head injury. The Executive Committee of the International Selfotel Trial. J Neurosurg. 2000 Jan;92(1):1-6. doi: 10.3171/jns.2000.92.1.0001. PMID 10616075
- [Background] Rosner MJ, Daughton S. Cerebral perfusion pressure management in head injury. J Trauma. 1990 Aug;30(8):933-40; discussion 940-1. doi: 10.1097/00005373-199008000-00001. PMID 2117669
- [Background] Gerber LM, Chiu YL, Carney N, Hartl R, Ghajar J. Marked reduction in mortality in patients with severe traumatic brain injury. J Neurosurg. 2013 Dec;119(6):1583-90. doi: 10.3171/2013.8.JNS13276. Epub 2013 Oct 8. PMID 24098983
- [Background] Farahvar A, Gerber LM, Chiu YL, Carney N, Hartl R, Ghajar J. Increased mortality in patients with severe traumatic brain injury treated without intracranial pressure monitoring. J Neurosurg. 2012 Oct;117(4):729-34. doi: 10.3171/2012.7.JNS111816. Epub 2012 Aug 17. PMID 22900846
- [Background] Rajajee V, Vanaman M, Fletcher JJ, Jacobs TL. Optic nerve ultrasound for the detection of raised intracranial pressure. Neurocrit Care. 2011 Dec;15(3):506-15. doi: 10.1007/s12028-011-9606-8. PMID 21769456
- [Background] Geeraerts T, Launey Y, Martin L, Pottecher J, Vigue B, Duranteau J, Benhamou D. Ultrasonography of the optic nerve sheath may be useful for detecting raised intracranial pressure after severe brain injury. Intensive Care Med. 2007 Oct;33(10):1704-11. doi: 10.1007/s00134-007-0797-6. Epub 2007 Aug 1. PMID 17668184
- [Background] Moretti R, Pizzi B. Optic nerve ultrasound for detection of intracranial hypertension in intracranial hemorrhage patients: confirmation of previous findings in a different patient population. J Neurosurg Anesthesiol. 2009 Jan;21(1):16-20. doi: 10.1097/ANA.0b013e318185996a. PMID 19098619
- [Background] Rajajee V, Fletcher JJ, Rochlen LR, Jacobs TL. Comparison of accuracy of optic nerve ultrasound for the detection of intracranial hypertension in the setting of acutely fluctuating vs stable intracranial pressure: post-hoc analysis of data from a prospective, blinded single center study. Crit Care. 2012 May 11;16(3):R79. doi: 10.1186/cc11336. PMID 22578001
- [Background] Hansen HC, Lagreze W, Krueger O, Helmke K. Dependence of the optic nerve sheath diameter on acutely applied subarachnoidal pressure - an experimental ultrasound study. Acta Ophthalmol. 2011 Sep;89(6):e528-32. doi: 10.1111/j.1755-3768.2011.02159.x. Epub 2011 Apr 21. PMID 21518306
- [Background] Hansen HC, Helmke K. Validation of the optic nerve sheath response to changing cerebrospinal fluid pressure: ultrasound findings during intrathecal infusion tests. J Neurosurg. 1997 Jul;87(1):34-40. doi: 10.3171/jns.1997.87.1.0034. PMID 9202262
- [Background] Dubourg J, Messerer M, Karakitsos D, Rajajee V, Antonsen E, Javouhey E, Cammarata A, Cotton M, Daniel RT, Denaro C, Douzinas E, Dubost C, Berhouma M, Kassai B, Rabilloud M, Gullo A, Hamlat A, Kouraklis G, Mannanici G, Marill K, Merceron S, Poularas J, Ristagno G, Noble V, Shah S, Kimberly H, Cammarata G, Moretti R, Geeraerts T. Individual patient data systematic review and meta-analysis of optic nerve sheath diameter ultrasonography for detecting raised intracranial pressure: protocol of the ONSD research group. Syst Rev. 2013 Aug 6;2:62. doi: 10.1186/2046-4053-2-62. PMID 23919384